CLINICAL TRIAL: NCT03830164
Title: Pentoxifylline, Atorvastatin, and Vitamin E (PAVE) as Treatment for Radiation-Induced Erectile Dysfunction
Brief Title: Pentoxifylline, Atorvastatin, and Vitamin E in Treating Patients With Erectile Dysfunction After Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0785; NCI-2019-00235 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0785 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Male Erectile Disorder; Prostate Adenocarcinoma; Erectile Dysfunction, CTCAE; Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Atorvastatin; Pentoxifylline; alpha-Tocopherol; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atorvastatin, vitamin E, pentoxifylline) (Experimental): Patients receive atorvastatin PO QD for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Beginning week 7, patients receive atorvastatin PO QD, vitamin E PO QD, and pentoxifylline PO TID for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atorvastatin; Drug: Pentoxifylline; Dietary Supplement: Vitamin E Compound

INTERVENTIONS:
Drug: Atorvastatin — Given PO
Drug: Pentoxifylline — Given PO
  Other Names: Oxpentifylline; Pentoxyphylline; PTX; Trental
Dietary Supplement: Vitamin E Compound — Given PO
  Other Names: 2,5,7,8-tetramethyl-2-(4,8,12-trimethyltridecyl)chroman-6-ol; E Vitamin; Vitamin E

SUMMARY:
This phase II trial studies how well pentoxifylline, atorvastatin, and vitamin E (PAVE) work in treating patients with erectile dysfunction after radiation therapy for prostate cancer. Atorvastatin may reduce high cholesterol. Pentoxifylline and vitamin E may enhance blood flow. Giving PAVE may work better in treating prostate cancer patients with post-radiation therapy erectile dysfunction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of patients who achieve a clinically significant improvement in erectile dysfunction (ED) when treated with a combination of atorvastatin or patient's currently prescribed statin, vitamin E, and pentoxifylline (PAVE).

SECONDARY OBJECTIVES:

I. To report the safety profile of PAVE. II. To report the rate of choosing other ED treatments after PAVE.

OUTLINE:

Patients receive atorvastatin orally (PO) once daily (QD) for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Beginning week 7, patients receive atorvastatin PO QD, vitamin E PO QD, and pentoxifylline PO thrice daily (TID) for up to 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* Previous radiation therapy (any form) with curative intent for prostate cancer
* Erectile dysfunction, as determined by an International Index of Erectile Function (IIEF)-5 score of < 22
* Normal testosterone (including men on testosterone replacement), defined as testosterone > 150 ng/dl at the time of screening
* Karnofsky Performance Status (KPS) >= 70, or Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients may be taking an HMG-coA-reductase inhibitor
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 X upper limits of normal (ULN)
* Creatinine kinase < 5 times ULN
* Normal renal function is defined as creatinine clearance >= 30 ml/min via the Cockcroft Gault formula

Exclusion Criteria:

* No androgen deprivation therapy within the past 12 months
* No contraindication to an HMG-coA-reductase inhibitor, vitamin E or pentoxifylline
* Not currently taking cyclosporine, the human immunodeficiency virus (HIV) protease inhibitors, hepatitis C protease inhibitors, gemfibrozil, other fibrates, clarithromycin, itraconazole or strong inhibitors of CYP3A4
* No recent cerebral or retinal hemorrhage that in the opinion of the treating physician would make PAVE unsafe (within 6 months)
* No current chemotherapy during study participation
* No active liver or muscle disease that in the opinion of the treating physician would make PAVE unsafe
* No prior radical prostatectomy, cystoprostatectomy, abdominoperineal resection or retroperitoneal lymph node dissection
* Not currently taking a 5PDE inhibitor nor have used one within 30 days of enrolling in the study
* No recent deep venous thrombosis, myocardial infarction or pulmonary embolism (within 6 months) requiring continued anticoagulation other than aspirin (acetylsalicylic acid [ASA])
* No cardiac arrhythmias or artificial heart valves requiring anticoagulation other than ASA
* No concurrent drugs with anti-platelet therapy properties (e.g., P2Y12 inhibitors, non-steroidal anti-inflammatory agents, selective serotonin reuptake inhibitors) other than low dose ASA (81 mg/d)
* Not currently taking high dose statin therapy, defined as rosuvastatin > 10 mg/d or atorvastatin > 40 mg/d
* Not currently taking theophylline
* No history of active peptic ulcer disease in the past 6 months
* No history of intolerance to pentoxifylline or methylxanthines such as caffeine, theophylline and theobromine that in the opinion of the treating physician would make PAVE unsafe
* No concurrent use of CYP1A2 inhibitors (e.g., ciprofloxacin), ketorolac, or vitamin K antagonists (e.g. warfarin)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: November 2019 to April of 2021. The recruitment of the participants occurred at the clinic and remotely via telephone calls.
Groups:
- Cohort 1: Participants not on any statin and were started on Atorvastatin 10 mg 1 tab daily with addition of receiving Pentoxyfilline 400 mg 1 tab 3 times daily and Vitamin E 1000units 1 tab daily.
- Cohort 2: Participants were on some amount of Atorvastatin and the dosage ramined the same With addition of receiving Pentoxyfilline 400 mg 1 tab 3 times daily and Vitamin E 1000units 1 tab daily.
- Cohort 3: Participants on some other statin beside atorvastatin and the dosage remained the same with addition of receiving Pentoxyfilline 400 mg 1 tab 3 times daily and Vitamin E 1000units 1 tab daily.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 5 | 8 | 1
Completed | 3 | 0 | 1
Not Completed | 2 | 8 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 5 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 5 | 8 | 1 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 1 | 9
  >=65 years | 1 | 4 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 8 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 8 | 0 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 4 | 6 | 1 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in International Index of Erectile Function (IIEF) Scores
Description: To estimate the proportion of participants who achieve a clinically significant improvement in erectile dysfunction (ED) when treated with a combination of Atorvastatin or participant's currently prescribed statin, Vitamin E, and Pentoxifylline (PAVE)
Time Frame: 12 months
Population: The data shows that 0 participants achieved any clinically significant improvement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 0 | 1
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Incidence of Adverse Events (AEs)
Description: The safety profile of the pentoxifylline, atorvastatin and vitamin E (PAVE) combination will be reported for each cohort, with adverse events summarized by grade and time to onset to first grade 3 adverse event.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 8 | 1
Participants
  Serious Adverse Event | 0 | 0 | 0
  Adverse Event | 0 | 2 | 0

3. Secondary Outcome: Choosing Other Erectile Dysfunction (ED) Treatments After Pentoxifylline, Atorvastatin and Vitamin E (PAVE)
Description: To report the rate of choosing other ED treatments after PAVE.
Time Frame: Up to 12 months
Population: No participants on cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 0 | 1
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: at baseline and throughout the trial and at 30 days after stopping the active treatment portion of this trial and the serious adverse events were captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdraws consent, up to 12 months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 0/5 | 2/8 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=8) | Cohort 3 (N=1)
Stomach Pain (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Blurry vision (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03830164/Prot_SAP_000.pdf